CLINICAL TRIAL: NCT02090244
Title: Förbättrar PTH Postero-lateral fusionsläkning Vid Ryggkirurgi?
Brief Title: Does PTH 1-34 (Teriparatide) Enhance Spinal Fusion in Humans?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Torsten Johansson, MD, PhD, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTH spinal stenosis; 2011-002917-12 (EudraCT Number)
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Spinal Stenosis
Keywords: PTH; Spinal stenosis; Teriparatide
MeSH Terms: conditions — Spinal Stenosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard care postoperatively.
- Teriparatide (Experimental): One injection daily for 4 weeks
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Daily injections with teriparatide 20 µg (PTH 1-34 (Forteo®)) during four weeks
  Other Names: Forteo
  Arms: Teriparatide

SUMMARY:
Parathyroid (PTH) hormone has been shown to enhance fracture healing in animal studies. There are so far only three published papers concerning humans. Postero-lateral fusions have shown a healing rate of less than 50% after bone. The purpose of this study is to determine if PTH 1-34 (teriparatide) improves the healing rate and the clinical course after spinal stenosis surgery.

DETAILED DESCRIPTION:
100 patients undergoing surgery due to spinal stenosis and intraoperatively treated with autologous bone graft, will be randomised to either 4 weeks of daily injections with teriparatide or control.

Primary outcome: The rate of healing at 6 months on CT Scans. Secondary outcomes; Pain (VAS), function (Oswestry Disability Index), quality of life (EQ-5D) at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* lumbar spinal stenosis operated on with decompression and bone grafting. All ages are accepted, but women must be postmenopausal.

Exclusion Criteria:

* •dementia or psychiatric disorder

  * known malignancy < 5 years prior to fracture
  * calcium above reference value
  * signs of liver disease
  * creatinine over ref. value
  * inflammatory joint disease
  * alcohol or drug abuse
  * oral corticosteroid medication
  * long-term NSAID-treatment (=> 3 months prior to fracture)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
The rate of bone healing after spinal stenosis surgery | 6 months + more than 2 years postoperatively.
  A radiologist, blinded to the treatment, will review all CT scans and judge whether there is a bony healing between the vertebrae.

SECONDARY OUTCOMES:
Pain | At 3 and 6 months.
  Pain is evaluated using VAS (Visual analogue scale). Zero means no pain and 10 is maximal pain.
Function | At 3 and 6 months.
  Function is evaluated using Oswestry Disability Index. Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Ottesen, MD, Principal Investigator — Ryggkliniken, US Linköping; Patrik Bernestrå, MD, Principal Investigator — Ortopedkliniken, Kalmar, Sweden
Locations (2):
- Sweden (2):
  - Ortopedkliniken, Kalmar
  - Ryggkliniken, US Linköping, Linköping